CLINICAL TRIAL: NCT02158260
Title: A New Method To Reduce Gastric Missing Areas in Capsule Endoscopy: a Single Center, Prospective and Self-controlled Trial
Brief Title: A New Method To Reduce Gastric Missing Areas in Capsule Endoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Side Liu, professor,MD,phD, Nanfang Hospital, Southern Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: capsule endoscopy20140107
Record Dates: First submitted 2014-05-31; First posted 2014-06-06 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Capsule Endoscopy
Keywords: Capsule endoscopy; Patient position changing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- position changing (Experimental): During the examination, subjects changed position in the following sequence: left lateral head-down position, supine position, prone head-down position, right lateral head-down position, supine position, left lateral position, prone position, prone hip-high position, right lateral position and sitting position.
  Interventions: Behavioral: Position changing
- free position (No Intervention)

INTERVENTIONS:
Behavioral: Position changing
  Arms: position changing

SUMMARY:
It is a single center, prospective and self-controlled trial. We'd like to explore a new method by changing position to reduce gastric missing areas in Capsule Endoscopy(CE)

DETAILED DESCRIPTION:
Background:Capsule endoscopy is widely used to observe small intestine.While it may miss important areas in stomach，especially in fundus.So far,physicians have no methods to observe stomach without no-missing areas by capsule endoscopy.

Objective:To explore a new method to reduce the areas missed by CE.

Methods:Subjects were prospectively enrolled.Every subjects will undergo 2 capsule endoscopies and 1 gastroscope.First capsule endoscopy,every subject have a better gastric preparation before swallowing CE and change position during the procedure.Second capsule endoscopy,every subject have a conventional CE. And then, every subject have a gastroscope.

Measurements:The primary measurements included safety, gastric preparation, visualization of gastric mucosa and rate of lesion detection.

ELIGIBILITY:
Inclusion Criteria:

* Subjects don't have swallowing difficulties, motility disorders, or a medical history that included abdominal surgery or obvious gastrointestinal strictures are included.

Exclusion Criteria:

* Subjects with swallowing difficulty, motility disorders, diabetes, life-threatening conditions, mental disorders, or patients that could be pregnant, have a cardiac pacemaker, electrical implant, or any other condition that would preclude compliance with the study requirements and/or device instructions are excluded from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
visualization of gastric mucosa | 1 year
  Gastric preparation included the degree of cleanliness and distention.Cleanliness was evaluated by 3 grades: good (the fluid was transparent and <5% of gastric mucosa was obscured by stomach contents), moderate (the fluid was a little opaque or 5% to 10% of gastric mucosa was obscured by stomach contents) and poor (the fluid was opaque or >10% of gastric mucosa was obscured by stomach contents). Distention was evaluated by 3 grades: good (existence of a small amount of gastric folds), moderate (existence of significant amount of gastric folds and gastric cavity was smaller than expected) and poor (gastric cavity was not inflated).

SECONDARY OUTCOMES:
rate of lesion detection | 1 year
  Gastroscope is the golden standard in diagnosing gastric diseases.we defined rate of lesion detection as the lesions detected by CE compared to gastroscope.

CONTACTS AND LOCATIONS:
Overall Officials: Side Liu, phD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China